CLINICAL TRIAL: NCT04985981
Title: The Prediction of Anastomotic Insufficiency Risk After Colorectal Surgery (PANIC) Study: Development and External Validation of an International, Multicenter Machine Learning Algorithm for Prediction of Anastomotic Insufficiency After Colonic or Colorectal Anastomosis
Brief Title: The Prediction of Anastomotic Insufficiency Risk After Colorectal Surgery (PANIC) Study
Status: Suspended | Type: Observational
Why Stopped: Change in core study organization
Sponsor: Michel Adamina, MD (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other); University Hospital, Geneva (Other); Clarunis - Universitäres Bauchzentrum Basel (Other); University Hospital, Basel, Switzerland (Other); University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Michel Adamina, MD, Chefarzt, Kantonsspital Winterthur KSW
Organization: Kantonsspital Winterthur KSW (Other)
Other Study IDs: PANIC
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Anastomotic Leak; Colorectal Cancer; Diverticulosis; Crohn Disease; Ulcerative Colitis; Mesenteric Ischemia
Keywords: Anastomotic Leak
MeSH Terms: conditions — Anastomotic Leak; Colorectal Neoplasms; Diverticulum; Crohn Disease; Colitis, Ulcerative; Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Prediction of Anastomotic Insufficiency risk after Colorectal surgery (PANIC) study aims to establish a machine-learning-based application that allows for accurate preoperative prediction of patients at risk for anastomotic insufficiency after colon and colorectal surgery.

DETAILED DESCRIPTION:
Anastomotic insufficiency leads to clinical strains for patients, and significantly increases morbidity and mortality. On average, hospital stay is extended by 12 days while healthcare-related expenses are increased by 30,000 USD when patients suffer from an anastomotic leak. In experienced centers, the approximated incidence of anastomotic insufficiency is 3,3% for colon and 8.6% for colorectal procedures. Multiple subgroups of patients with increased risk for anastomotic leaks have been described in previous publications. Meticulous preoperative recognition of patients with increased risk for anastomotic insufficiency is clinically beneficial, as it would permit improved ressource preparation, enhanced patient education and superior surgical decision-making. However, it is often difficult for clinicians to balance the plethora of crucial risk factors for anastomotic leaks for a single patient. Machine learning methods have been exceptionally effective at incorporating various clinical variables into one unified risk prediction model. To the authors' best knowledge, there does not yet exist a credible prediction model or a conclusive prediction score for anastomotic insufficiency after colon and colorectal anastomosis. The aim of the Prediction of Anastomotic Insufficiency risk after Colorectal surgery (PANIC) study is to establish and externally validate an efficient machine-learning-based prediction tool based on multicenter data from a range of international centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent colon or colorectal anastomosis for neoplasia, diverticulitis, mesenterial ischemia, iatrogenic or traumatic perforation, or inflammatory bowel disease

Exclusion Criteria:

* age < 18
* recurrent colorectal cancer
* peritoneal carcinomatosis or unresectable metastatic disease at time of bowel resection
* informed consent not obtainable
* follow-up < 6 weeks after surgery
* no reversal of and ostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent colon or colorectal anastomosis for neoplasia, diverticulitis, mesenterial ischemia, iatrogenic or traumatic perforation, or inflammatory bowel disease. Only patients who have reached the age of 18 will be accepted. Only patients who are able to give informed consent to the procedure will be accepted.
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Anastomotic leak | 5 years
  Occurrence of anastomotic insufficiency/leak is defined as any clinical signs of leakage, confirmed by radiological examination, endoscopy, clinical examination of the anastomosis, or upon reoperation.

SECONDARY OUTCOMES:
Occurrence of Death | 90 days
Time to diagnosis of anastomotic leak | 90 days
  Time to diagnosis of a leakage will be calculated as days between the index operation and diagnosis of the leakage by imaging with extraluminal contrast, endoscopy, re-operation, or when fecal containing fluid is objectified in a drainage.

OTHER OUTCOMES:
Disease-free survival (months) | 5 years
Overall survival (months) | 5 years
Adjuvant/additive immunochemotherapy (yes/no) | 5 years
  Did the patient receive adjuvant/additive immunochemotherapy after surgery? (yes/no)
Adjuvant/additive radiotherapy (yes/no) | 5 years
  Did the patient receive adjuvant/additive radiotherapy after surgery? (yes/no)
Additive curative surgery (no/yes: liver; lung; locoragional relapse) | 5 years
  Did the patient receive additive curative surgery after the initial intervention? (no/yes: liver; lung; locoragional relapse)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Adamina, Prof. Dr. med., Study Chair — Clinical Research and Artificial Intelligence in Surgery, Department of Biomedical Engineering, University of Basel, Allschwil, Switzerland; Anas Taha, Dr. med., Principal Investigator — None currently; Thomas Steffen, Principal Investigator — Cantonal Hospital of St. Gallen; Stephanie Taha-Mehlitz, Dr. med., Principal Investigator — Department of Visceral Surgery, Clarunis, University Hospital Basel, Basel, Switzerland; Frédéric Ris, Prof. Dr. med., Principal Investigator — Department of Surgery, Hôpitaux Universitaires de Genève
Locations (2):
- Switzerland (2):
  - Clinical Research and Artificial Intelligence in Surgery, Department of Biomedical Engineering, University of Basel, Allschwil, Switzerland, Allschwil, Basel
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2020-12-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT04985981/Prot_001.pdf